CLINICAL TRIAL: NCT07140042
Title: Comparison of Physical Fitness, Physical Activity Level, Depression and Quality of Life in Bipolar and Schizophrenia Patients With Healthy Controls
Brief Title: Physical Fitness, Physical Activity Level, Depression and Quality of Life in Bipolar and Schizophrenia Patients
Status: Completed | Type: Observational
Sponsor: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İsmail Koç, Assist Prof, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Other Study IDs: IKoc
Record Dates: First submitted 2025-07-22; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-07

CONDITIONS: Bipolar Disorder (BD); Schizophrenia Disorder
MeSH Terms: conditions — Bipolar Disorder; Schizophrenia | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Bipolar group: Bipolar disorder
  Interventions: Other: Survey
- schizophrenia group: schizophrenia disorder
  Interventions: Other: Survey
- healthy control group: healthy control
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
Assessment of physical activity levels, physical fitness and quality of life of bipolar and schizophrenia patients is necessary to verify the effectiveness of treatments and care activities in Community Mental Health Centers (CMHCs) and to plan new therapeutic and rehabilitative activities. In one study, they found that physical activity level-physical fitness has a positive impact on psychiatric services and can improve physical health outcomes of patients with schizophrenia. They also found an improvement in psychological and social outcomes in these patients. Therefore, physical activity level and physical fitness are stated as critical parameters of biopsychosocial approach in mental health services.

The aim of this study was to compare physical fitness, physical activity level, depression and quality of life in bipolar and schizophrenia patients with healthy individuals.

DETAILED DESCRIPTION:
Bipolar disorder ranks among the top 20 causes of disability among all medical conditions worldwide and 6th among mental disorders. Bipolar disorder is defined as a serious mental illness involving emotional ups and downs. It is a disorder characterized by two distinct periods of illness, manic and depressive . These two periods of illness are characterized by remission and exacerbation. The patient completely returns to normal except for the periods of illness. The mania or outburst period is when the mood is very high. Bipolar patients have a reduced life expectancy and a higher risk of developing metabolic syndromes. It is a serious mental health problem in terms of mortality, morbidity and suicide . Bipolar individuals have a higher mortality and morbidity rate than the general population. Exercise and physical activity are highly effective in preventing mortality and cardiovascular diseases and can reduce the risk of cardiovascular disease. The International Organization of Physiotherapists recommends that individuals with mental illness should do at least 150 minutes of brisk walking or 75 minutes of physical activity per week.

Exercise is also an effective method in the treatment of mood disorders in patients with bipolar disorder. Aerobic physical exercises are also a good treatment for neurocognitive dysfunction in patients with bipolar disorder. Decreased walking capacity in hospitalized patients with bipolar disorder is due to impaired muscle conditioning, which affects daily living functions. At the same time, bipolar individuals have poorer exercise habits such as less walking and less strength exercises than healthy individuals. A qualitative study in bipolar patients also found that mood influences physical activity. Schizophrenia is a chronic mental disorder characterized by the occurrence of both positive symptoms such as hallucinations and delusions and negative symptoms such as apathy and withdrawal, repetition of cognitive skills and disorganization. Patients with schizophrenia have been found to be less physically active and less physically fit than the general population. Exercise is a subset of physical activity that is planned, structured and repetitive bodily movements performed to increase and maintain one or more parts of physical fitness.

Therefore, physical activity level and physical fitness are stated as critical parameters of biopsychosocial approach in mental health services.

The aim of this study was to compare physical fitness, physical activity level, depression and quality of life in bipolar and schizophrenia patients with healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* - Individuals diagnosed with bipolar and schizophrenia by a physician according to DSM-5 criteria
* Individuals with bipolar and schizophrenia between the ages of 18-64
* Patients without other concomitant psychiatric disorders
* Patients who can communicate
* Patients who agreed to participate in this study and gave informed consent

Exclusion Criteria:

* - Patients with a psychiatric diagnosis other than bipolar and schizophrenia. Pregnancy Not giving consent to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: bipolar and schizophrenia
Sampling Method: Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2025-06-23 (Actual); Primary Completion 2025-08-05 (Actual); Study Completion 2025-08-12 (Actual)

PRIMARY OUTCOMES:
Antropometric measurement | 2 week
  Antropometric measurement will be evaluated like weight, height, body mass index, circumferences etc.
International Physical Activity Questionnaire | 2 weeks
  To measure Physical Activity Level
Beck Depression Inventory | 2 weeks
  Depression
Short form 36 | 2 weeks
  Quality of life

CONTACTS AND LOCATIONS:
Locations (1):
- Yeditepe university, Istanbul, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No